CLINICAL TRIAL: NCT06341920
Title: BoneFit: A Student-led Multimodal Prehabilitation Service for Orthopaedic Surgical Patients in Hull
Brief Title: BoneFit: Multimodal Prehabilitation for People Preparing for Orthopaedic Surgery
Acronym: BoneFit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS198 - 332551
Record Dates: First submitted 2024-03-05; First posted 2024-04-02 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Orthopedic Disorder
Keywords: prehabilitation; optimisation; surgery; surgical preparation
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Intervention v control
Masking Description: Masking is not possible - referrals/care providers know whether they/referral is involved in the intervention or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BoneFit intervention (Experimental): Participants will receive a personalised care plan comprising exercise, nutrition and psychological wellbeing based on individual need in the 8-week period prior to surgery
  Interventions: Behavioral: Experimental: BoneFit intervention
- Control (Placebo Comparator): Participants who are allocated to this group will receive baseline tests and will be invited to re-attend 3 months post surgery to re-do tests. This group will receive usual care (no intervention). The groups will be compared.
  Interventions: Behavioral: Placebo Comparator: Control

INTERVENTIONS:
Behavioral: Experimental: BoneFit intervention — Exercise, nutrition and psychological support provided in 8 weeks prior to surgery
  Arms: BoneFit intervention
Behavioral: Placebo Comparator: Control — Control group receive usual care (zero intervention)
  Arms: Control

SUMMARY:
To conduct a pilot feasibility study to determine the effect of a student-led prehabilitation service in people awaiting total hip or knee replacement surgery.

DETAILED DESCRIPTION:
The aim of BoneFit is to provide local people living in the Hull region with a needs-based prehabilitation care package to improve their physical and mental health, quality of life & reduce their length of hospital stay, complications and readmission rates to hospital following orthopaedic surgery (total hip replacement, or total knee replacement.

Currently, Hull University Teaching Hospitals do not offer a prehabilitation service for local patients. The University of Hull will partner with them to provide a student-led multimodal prehabilitation service for referred patients awaiting orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Waiting for unilateral total hip or knee replacement surgery for a minimum of 6 months;
* Able to provide informed consent;

Exclusion Criteria:

* Previous hip or knee surgery;
* Any medical conditions for which moderate to vigorous exercise is contraindicated;
* Patellar or hip joint instability;
* Any other disease/condition which severely effects functional performance e.g. stroke or Parkinson's disease;
* Chronic depression or significant psychiatric disorder;
* Enrolled in a clinical trial (or recently completed one);
* Cognitive impairment which would affect compliance to BoneFIt service;
* Patients unable or unwilling to commit to required study follow-ups
* Pregnancy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 2 years
  Number of people recruited and trained
Adherence and attendance | 2.5 years
  Record the number of sessions attended and calculate adherence to protocol (%)
Acceptability | 3 years
  Conduct semi-structured interviews following the intervention with sample of participants and ask them about experiences of the intervention. The post-intervention interviews will focus on how participants viewed the intervention, perceived burdens, and perceived effectiveness from initiation through to completion. A list of burdens / perceived benefits will be reported alongside percentage rates of respondents.

SECONDARY OUTCOMES:
Physical fitness | 3 years
  Compare incremental shuttle walk test scores (intervention v controls). Units: stage achieved and time taken (seconds)
Length of stay | 3 years
  Compare days in hospital following surgery (intervention v controls). Units: hours in hospital following surgery.
Readmission rates | 3 years
  Compare the % of patients in each group who were readmitted to hospital following surgery (intervention v controls)
Overall quality of life | 3 years
  Compare quality of life scores (intervention v controls) using EQ-5D-5L questionnaire. Index scores range between zero and one, based on 5-point Likert scale, with scores closer to one indicating an improved status.
Knee or hip specific pain, function and quality of life | 3 years
  Compare knee or hip specific quality of life scores (intervention v controls). For knee replacements, the KOOS-12 is scored between 0-100 on 5-point Likert scale, with higher scores equating to improved status. For hip replacements, HOOS-12 scores between 0 to 4 points with 0 representing no hip problems and 4 representing extreme hip problems, based on response to 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ingle, Principal Investigator — Professor of Exercise Science for Health and Rehabiliation
Locations (1):
- Hull University Teaching Hospitals, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Please contact the PI and request access to data
Supporting Information: Study Protocol
Time Frame: Dec 2027
Access Criteria: Request from PI

REFERENCES:
- [Derived] Ingle L, Snook J, Smith L, Oliver B, Bray J, Wells L, Moorhouse J, Dixon L, Simpson P, Osman S, Saxton J, Rajendran A, Gopalakrishnan G, Symes T. Optimisation of the preparation phase for orthopaedic surgery: Study protocol for a student-led multimodal prehabilitation feasibility trial (BoneFit). PLoS One. 2025 Feb 12;20(2):e0314680. doi: 10.1371/journal.pone.0314680. eCollection 2025. PMID 39937759

DOCUMENTS (1):
  • Study Protocol (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT06341920/Prot_000.pdf